CLINICAL TRIAL: NCT01087268
Title: Randomized Double-Blind Controlled Phase III Trial of Hyperbaric Oxygen Therapy in Patients Suffering Long-Term Adverse Effects of Radiotherapy for Pelvic Cancer (HOT II)
Brief Title: Hyperbaric Oxygen Therapy in Treating Long-Term Gastrointestinal Adverse Effects Caused by Radiation Therapy in Patients With Pelvic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000667367; RMH-CCR3086; EUDRACT-2008-002152-26; EU-21010; MREC-08/H0903/40
Record Dates: First submitted 2010-03-13; First posted 2010-03-16 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2010-03

CONDITIONS: Bladder Cancer; Cervical Cancer; Colorectal Cancer; Endometrial Cancer; Gastrointestinal Complications; Long-term Effects Secondary to Cancer Therapy in Adults; Ovarian Cancer; Prostate Cancer; Radiation Toxicity; Sarcoma; Testicular Germ Cell Tumor; Vaginal Cancer
Keywords: gastrointestinal complications; radiation toxicity; long-term effects secondary to cancer therapy in adults; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; stage I bladder cancer; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage I vaginal cancer; stage II vaginal cancer; stage III vaginal cancer; stage I malignant testicular germ cell tumor; stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; stage I endometrial carcinoma; stage II endometrial carcinoma; stage III endometrial carcinoma; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IA ovarian epithelial cancer; stage IB ovarian epithelial cancer; stage IC ovarian epithelial cancer; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IA ovarian germ cell tumor; stage IB ovarian germ cell tumor; stage IC ovarian germ cell tumor; stage IIA ovarian germ cell tumor; stage IIB ovarian germ cell tumor; stage IIC ovarian germ cell tumor; stage IIIA ovarian germ cell tumor; stage IIIB ovarian germ cell tumor; stage IIIC ovarian germ cell tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Radiation Injuries; Sarcoma; Testicular Germ Cell Tumor; Vaginal Neoplasms; Rectal Neoplasms; Testicular Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Other: questionnaire administration
Procedure: gastrointestinal complications management/prevention
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Radiation therapy can cause long-term adverse effects. Hyperbaric oxygen therapy may be effective in lessening gastrointestinal symptoms caused by radiation therapy given for pelvic cancer. It is not yet known whether high-pressure oxygen is effective in treating adverse effects caused by radiation therapy.

PURPOSE: This randomized phase III trial is studying hyperbaric oxygen therapy to see how well it works in treating long-term gastrointestinal adverse effects caused by radiation therapy in patients with pelvic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the clinical benefits of hyperbaric oxygen therapy in reducing dysfunction in patients with pelvic cancer developing iatrogenic gastrointestinal symptoms as a result of previous radical pelvic radiotherapy completed at least one year ago.

OUTLINE: This is a multicenter study. Patients are stratified according to center and severity of symptoms (low vs high). Patients are randomized to 1 of 2 treatment arms.

* Arm I (treatment group): Patients undergo hyperbaric oxygen therapy over 90 minutes, 5 days a week, for 8 weeks for a total of 40 treatments. Oxygen at 100% is breathed for 30 minutes, followed by a 5-minute "air break" and a further 30 minutes of breathing oxygen. A further 5-minute "air break" is followed by a further 30 minutes of breathing oxygen. During the final 10 minutes of oxygen breathing, the chamber is depressurized to ambient atmospheric pressure at a linear rate (14.2 kPa/min).
* Arm II (control group): Patients undergo hyperbaric oxygen therapy over 90 minutes, 5 days a week, for 8 weeks for a total of 40 treatments. Oxygen at 21% is breathed for 30 minutes, followed by a 5-minute "air break" and a further 30 minutes of breathing oxygen. A further 5-minute "air break" is followed by a further 30 minutes of breathing oxygen. During the final 10 minutes of oxygen breathing, the chamber is depressurized to ambient atmospheric pressure at a linear rate (3 kPa/min).

Tissue samples from rectal biopsies may be collected and analyzed.

Patients complete questionnaires (Health Economics, Inflammatory Bowel Disease Questionnaire [IBDQ], EORTC Quality of Life [QLQ]-C30, and QLQ-CR38) at baseline and then at 3, 6, 9, and 12 months after the start of treatment.

After completion of study treatment, patients are followed within 14 days and at 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Past history of rectal, prostate, testicular, bladder, uterine cervix, uterine corpus, vaginal, or ovarian cancer

  * Malignant disease (T1-3, N0-1, M0)
* No evidence of cancer recurrence
* Gastrointestinal symptoms attributable to prior radiotherapy received at least 1 year ago, meeting 1 of the following criteria:

  * Grade 2 or higher in any Late Effects in Normal Tissues Subjective, Objective, Management, and Analytic Scales (LENT SOMA) category
  * Grade 1 with difficult intermittent symptoms
* Symptoms are not relieved by appropriate life-style advice and medication over a 3-month period

PATIENT CHARACTERISTICS:

* Must be physically and psychologically fit to undergo hyperbaric oxygen therapy
* No claustrophobia
* No epilepsy
* No chronic obstructive airway disease, bullous lung disease, acute or chronic pulmonary infection, uncontrolled asthma, or untreated pneumothorax
* No previous middle/inner ear operations (except grommets and similar procedures) and/or inability to equalize middle ear pressure
* No contraindication or other inability to undergo magnetic resonance imaging, if required to rule out malignancy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior surgery for rectal cancer
* No prior hyperbaric oxygen therapy (excluding treatment for decompression illness)
* No prior treatment with bleomycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms score using the IBDQ quality-of-life questionnaire

SECONDARY OUTCOMES:
Physician assessment of adverse effects using LENT SOMA scales of radiation injury
Patient self-assessments using EORTC QLQ-C30 and Defecation Problem Subscale of QLQ-CR38
Photographic images of rectal mucosa
Physician assessment of rectal dysfunction based on the modified CTCAE grading system
Health economics data

CONTACTS AND LOCATIONS:
Overall Officials: John R. Yarnold, MD, FRCR, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom